CLINICAL TRIAL: NCT06733090
Title: The Effect of Two Different Oral Care Solutions on the Prevention of Ventilator-associated Pneumonia in the Intensive Care Unit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MELEK UNLUGEDIK (Other)
Responsible Party: Sponsor-Investigator, MELEK UNLUGEDIK, Istanbul University - Cerrahpasa (IUC), Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0382
Record Dates: First submitted 2024-12-03; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Intensive Care Patients; Oral Care Performance; Intensive Care Nurses
Keywords: intensive care; oral care; oral care performance

STUDY DESIGN:
Intervention Model Description: The study will be conducted in two stages. In the first stage; Nurse Information Form and Ventilator Associated Pneumonia Knowledge pretest will be applied to nurses who accept to participate in the study before the training. A 2-week training program will be applied to nurses by the researcher. In the second stage of the study, the forms in the second stage will be applied to patients who meet the criteria for inclusion in the study and the process will be followed in the same way in two separate groups. According to the research sample calculation, it is planned to include at least 25 patients in the experimental group and 25 patients in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.2% chlorhexidine glucanate solution (Experimental): 0.2% chlorhexidine glucanate solution
  Interventions: Drug: 0.2% chlorhexidine glucanate solution
- 0.12% chlorhexidine glucanate solution (Experimental): 0.12% chlorhexidine glucanate solution
  Interventions: Drug: 0.12% chlorhexidine glucanate solution

INTERVENTIONS:
Drug: 0.12% chlorhexidine glucanate solution — The superiority of two different solutions over each other will be examined with a standard maintenance.
  Arms: 0.12% chlorhexidine glucanate solution
Drug: 0.2% chlorhexidine glucanate solution — 0.2% chlorhexidine glucanate solution
  Arms: 0.2% chlorhexidine glucanate solution

SUMMARY:
Ventilator-associated pneumonia (VAP) is a lung parenchymal tissue infection that develops nosocomially 48-72 hours after the start of mechanical ventilation (8, 15, 17, 23, 31). The second most common nosocomial infection in intensive care units in the United States is VAP (20). Approximately 90% of pneumonias developing in intensive care units are seen in patients receiving mechanical ventilation support, while the risk of VAP development is higher in the first days of hospitalization, and has been reported to be 3%/day in the first 5 days, 2%/day on the following six and ten days, and 1%/day on subsequent days (7, 20, 23,37). The concept of the Bundle of Care was first defined by the Institute for Healthcare Improvement in 2005 (21, 25). The Bundle of Care; It is a set of practices that have been beneficial in terms of clinical improvement, each of which includes 3-5 evidence-based, preventive interventions that contribute to the quality of care (5, 21, 25, 26, 30). There are studies in the literature showing that the use of the Care Bundle for the development of VAP reduces the rate of VAP development (5, 30, 34, 29, 28).

Evidence-based practices frequently recommended in the literature within the scope of the VAP Care Bundle are; giving the patient a semi-fowler position (sitting at a 30-45 degree angle), evaluating daily extubation, evaluating daily sedation, peptic ulcer prophylaxis unless contraindicated, and deep vein thrombosis prophylaxis (15, 21, 23, 26, 28, 30).

Health Care Improvement Institute; recommends washing hands before and after patient contact, removing subglottic secretions, and not changing ventilator circuits earlier than 48 hours (19, 21, 32, 33). In addition to evidence-based practices, the Institute for Health Care Improvement recommends that oral intubation be preferred to nasotracheal intubation, endotracheal tube cuff pressure should be between 20-30 cmH2O, enteral feeding should be initiated within 24-48 hours for hemodynamically stable intensive care patients, oral care should be performed with an antiseptic solution at 2-12 hour intervals, including teeth, cheeks, and tongue, monitoring humidifier filters and irrigation solutions, and aspiration should be performed under appropriate conditions. These interventions are considered evidence-based (1, 2, 3, 8, 9, 10, 11, 12, 14, 16, 18, 22, 23, 26, 33).

The evidence-based Care Bundle Interventions to be implemented by the researcher within the scope of this study are listed below. Interventions to be implemented by the nurse's decision include; Oral care with 0.12% chlorhexidine glucanate or 0.2% chlorhexidine glucanate solution, 4 times a day, at 6-hour intervals, semi-fowler position (sitting at a 30-45 degree angle) unless contraindicated, monitoring the endotracheal tube cuff pressure to be between 20-30 cmH2O, changing ventilator circuits and humidifier filters in case of visible contamination or malfunction, and monitoring the aspiration application. Interventions to be implemented by the physician's decision include; includes daily extubation assessment, peptic ulcer prophylaxis unless contraindicated, deep vein thrombosis prophylaxis unless contraindicated.

DETAILED DESCRIPTION:
The study was planned to examine the effects of two different solutions (0.12% chlorhexidine glucanate and 0.2% chlorhexidine glucanate) on the incidence of VAP in patients who receive the VAP Care Bundle, which was created with evidence-based practices recommended in the literature, after the training to be given to nurses who provide care to patients on mechanical ventilation in the General Intensive Care Unit.

The study will be conducted in 2 stages. The first stage, in which nurses working in the Intensive Care Unit will be included in the sample group; was planned in a pretest-posttest design, in a single group, in order to determine the effectiveness of the training to be applied to the nurses.

The research will be conducted in two stages. The first stage, in which nurses working in the Intensive Care Unit will be included in the sample group, was planned in a pretest-posttest design, in a single group, in order to determine the effectiveness of the training to be given to nurses. The second stage was planned in a single-group, prospective experimental design, in order to determine the effect of the VİP Care Bundle application on the VİP incidence and the duration of stay on the ventilator. In the first stage of the research that nurses working in the General Intensive Care Unit of the Republic of Turkey Ministry of Health Silivri State Hospital will constitute the universe of the study. Those of these nurses who meet the inclusion criteria will be included in the sample group.

It will be conducted in the General Intensive Care Unit of the Republic of Turkey Ministry of Health Istanbul Silivri State Hospital. There are a total of 9 patient beds in the institution where the study will be implemented. The unit is a Level 3 intensive care unit. There are 20 nurses working in this unit. Nurse Information Form, Ventilator-Associated Pneumonia Information Test will be used.

In the second stage; after the completion of the nurse education program, patients who meet the inclusion criteria that will be grouped with simple randomization; Patient Information Form will be filled in on the day the patient is connected to the ventilator in the intensive care unit, VAP Prevention Protocol Monitoring Form and GKS (Glasgow Coma Scale) for each day the patient is connected to the ventilator, APACHE II (Acute Physiology and Chronic Health Evaluation II) 24 hours after the patient is admitted to the unit, and CPIS (Clinical Pulmonary Infection Score) will be filled in on the 1st, 3rd, and 5th hospitalization days following the patient's connection to the ventilator. At this stage, the oral health of the patients will be evaluated with the Oral Health Evaluation Form (permission was obtained from Assoc. Prof. Dr. Aylin Palloş via e-mail.). 0.12% chlorhexidine glucanate solution or 0.2% chlorhexidine glucanate solution will be used as oral care solution. The solutions are registered in the Product Tracking System of the Ministry of Health, Turkish Medicines and Medical Devices Agency. Oral care practices of the patients will be carried out in accordance with the Appendix 8. Special Oral Care Protocol, which was created by reviewing the literature (39,40). Oral care practices will be carried out by the researcher between 08:00-17:00 since the researcher is actively working in this intensive care unit. Oral care practices between 17:00-08:00 will be carried out by the nurse who has been trained and works in the night shift. The Information Form will be filled in by the researcher, the VAP Prevention Protocol Follow-up Form, the Oral Health Evaluation Form will be filled in by the nurses who provide care to the patient (The researcher is actively working in this intensive care unit), the GKS (Glasgow Coma Scale) will be filled in from the nurses' notes, the APACHE II (Acute Physiology and Chronic Health Evaluation II) will be filled in from the patient records (Institutional permission has been obtained), and the CPIS (Clinical Pulmonary Infection Score) will be filled in by the physician. The GKS (Glasgow Coma Scale) and APACHE II (Acute Physiology and Chronic Health Evaluation II) forms are routinely filled in the unit where the study is conducted for the patients in the sample group. The Oral Health Assessment Form will be filled in daily (24-hour intervals) after 4 applications for each patient, starting with the first assessment at admission, until the patient is discharged. The data obtained as a result of the study will be evaluated with appropriate statistical methods. In addition, the incidence of ventilator-associated pneumonia obtained at the end of the study will be compared with the data recorded by the Infection Control Committee for the General Intensive Care Unit and recorded in the Ministry of Health system. These dates correspond to 1 year before the period in which the research data were collected.

The second stage; 0.12% chlorhexidine glucanate solution or 0.2% chlorhexidine glucanate solution will be used in oral care with the standard VAP Care Bundle application. The group to which the patients will be included will be determined by the nurse in charge of the service through simple randomization. This study was planned in a two-group, prospective, experimental design to determine the effect of oral care intervention applied with two different solutions on the prevention of ventilator-associated pneumonia.

It was planned to examine the effect of two different solutions (0.12% chlorhexidine glucanate and 0.2% chlorhexidine glucanate) on the incidence of VAP in patients who used the VAP Care Bundle, which was created with evidence-based practices recommended in the literature, after the training to be given.

The research will be carried out in 2 stages. The first stage, in which nurses working in the Intensive Care Unit will be included in the sample group; It was planned in a pretest-posttest design, in a single group, in order to determine the effectiveness of the training to be applied to the nurses.

The second stage; 0.12% chlorhexidine glucanate solution or 0.2% chlorhexidine glucanate solution will be used in oral care with the standard VAP Care Bundle application. The group in which the patients will be included will be determined by the responsible nurse of the service through simple randomization. This study was planned as a two-group, prospective, experimental design to determine the effect of oral care intervention applied with two different solutions on the prevention of ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

Invasive mechanical ventilation support (at least 48 hours) 18 years of age or older Obtaining the approval of the legal guardian for his/her care

Exclusion Criteria:

Chronically dependent on a ventilator Chlorhexidine gluconate sensitivity Diagnosed with VAP before the data collection process Semi-fawler position not applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
APACHE II (Acute Physiology and Chronic Health Evalution II | It is filled only once for each patient, at the end of the 24th hour.
  Patients will be examined immediately after 24 hours after being admitted to intensive care. It will be looked at once.
Follow-up period of patients checklist | If ex or not discharged, the longest period is determined as 30 days.
  It indicates how long patients will be followed. Patients are followed until they are discharged from intensive care and until they die. If ex or not discharged, the longest period is determined as 30 days.
CPIS Clinical Pulmonary Infection Score | It is filled out once for the 1st, 3rd and 5th days when the patient is admitted to the intensive care unit.
  CPIS (Clinical Pulmonary Infection Score) will be filled in on the 1st, 3rd and 5th hospital days.
GKS Glasgow Coma Scale | once a day on the day the patient is admitted to the intensive care unit, for a maximum of 30 days until death or discharge, whichever came first
  GKS Glasgow Coma Scale, It will be checked once a day every day. It is a method that aims to record a person's state of consciousness reliably and objectively at the beginning and in subsequent evaluations. When the patient is evaluated according to the criteria of the scale, the patient is given scores between 3 (indicating profound loss of consciousness) and 14 (according to the original scale) or 15 (according to the widely used corrected scale).
Oral Health Evaluation Form | once a day on the day the patient is admitted to the intensive care unit, for a maximum of 30 days until death or discharge, whichever came first
  The oral health of the patients will be checked once a day by the researcher from the first moment throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Avcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I am the principal investigator and contact person.